CLINICAL TRIAL: NCT00833222
Title: Neuroendocrine Mechanisms of Growth and Body Composition in Preterm and Term Infants
Acronym: PREMA
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Other Study IDs: 24087
Record Dates: First submitted 2009-01-29; First posted 2009-02-02 (Estimated); Last update posted 2017-12-26 (Actual); Status verified 2017-12

CONDITIONS: Premature Birth
Keywords: premature birth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva; Urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Full Term Infants: Infants born between 37 4/7 weeks and 42 3/7 weeks gestation.
- Preterm Infants: Infants born between 32 4/7 weeks and 35 3/7 weeks gestation.

SUMMARY:
The purpose of this study is to test the feasibility of measuring body composition by air displacement plethysmography (ADP) in rapidly growing, medically stable late gestation [32-35 weeks post-menstrual age (PMA)] premature infants.

DETAILED DESCRIPTION:
1. To assess the feasibility of measuring body fat deposition by ADP in medically stable late gestation (32-35 weeks), premature infants during a period of rapid postnatal growth.
2. To test the relationship between %BF by ADP to %BF by DXA, as well as characterize the relationship between these fat measures with bone measures by quantitative ultrasound and serum levels of insulin, IGF-1, IGF binding proteins, adiponectin and leptin.
3. To perform inter- and intra-rater testing of anthropometric, ultrasound, and ADP measurements.
4. Compare growth, body composition and bone strength between infants born preterm to infants born full term.

ELIGIBILITY:
Inclusion Criteria:

* Infants born between 32 4/7 and 35 3/7 weeks gestation or 37 4/7 and 42 3/7 weeks gestation, by physical exam at birth
* Birth weight between the 5th and 95th percentile corrected for gestational age

Exclusion Criteria:

* Chromosomal abnormalities
* Major congenital anomalies
* Major surgery
* Severe CNS injury
* Inborn errors of metabolism
* Assisted ventilation
* Inability to start enteral feeds by 96 hours of age

Ages: 31 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Premature and full term infants admitted to the University of Utah Newborn Intensive Care Unit, Intermediate Nursery or Well Baby Nursery
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2008-01; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Growth trajectory | Weekly

CONTACTS AND LOCATIONS:
Overall Officials: Laurie Moyer-Mileur, PhD, Principal Investigator — University of Utah; Kristine Jordan, MPH, PhD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States